CLINICAL TRIAL: NCT00004081
Title: A Phase II Trial of Weekly, Low-Dose Docetaxel (Taxotere) in Patients With Platinum-Resistant Epithelial Ovarian or Primary Peritoneal Serous Cancer
Brief Title: Docetaxel in Treating Women With Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Cannistra, MD, Investigator, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067292; BIH-99-1286; NCI-V99-1565
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating women who have ovarian epithelial cancer or primary peritoneal cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of docetaxel in women with platinum resistant, refractory ovarian epithelial or primary peritoneal serous cancer.

OUTLINE: Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive a minimum of 6 courses of therapy, including 2 courses beyond CR.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal serous cancer that is resistant to platinum therapy
* Platinum resistance as defined by one of the following:

  * Relapse within 6 months of platinum based chemotherapy
  * Residual disease after completion of platinum based chemotherapy
  * Disease progression while receiving platinum based chemotherapy
  * Marker only relapse (CA-125 elevation) and measurable disease
* Bidimensionally measurable disease on exam or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 2 months

Hematopoietic:

* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGPT or SGOT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* Acceptable cardiac exam
* No active cardiac ischemia

Pulmonary:

* Acceptable pulmonary exam
* No active pulmonary infection or compromise

Other:

* Not pregnant or nursing
* No severe peripheral neuropathy (grade 2 or greater)
* No other significant psychiatric or medical conditions that would interfere with compliance
* No other malignancies within the past 3 years, except:

  * Limited basal or squamous cell skin cancer
  * Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior cytokine therapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for ovarian epithelial or peritoneal serous cancer
* Prior paclitaxel allowed
* No prior docetaxel
* At least 3 years since prior chemotherapy for other disease

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior pelvic radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-07; Primary Completion 2002-01 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Cannistra, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Berkenblit A, Seiden MV, Matulonis UA, Penson RT, Krasner CN, Roche M, Mezzetti L, Atkinson T, Cannistra SA. A phase II trial of weekly docetaxel in patients with platinum-resistant epithelial ovarian, primary peritoneal serous cancer, or fallopian tube cancer. Gynecol Oncol. 2004 Dec;95(3):624-31. doi: 10.1016/j.ygyno.2004.08.028. PMID 15581974